CLINICAL TRIAL: NCT01047631
Title: Relationship of Cardiovascular and Muscular Capacity to Daily Functioning in Frail Older Adults
Brief Title: Role of Exercise in Diastolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Neil Alexander, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1997-585
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2010-01

CONDITIONS: Diastolic Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional circuit training and lifestyle counseling (Experimental)
  Interventions: Behavioral: Functional circuit training and lifestyle counseling
- Health education and independent walking (Active Comparator)
  Interventions: Behavioral: Health education and independent walking

INTERVENTIONS:
Behavioral: Functional circuit training and lifestyle counseling — Tests are performed at the beginning, and repeated after 12 and 24 weeks:
  * Measure general fitness levels such as walking, strength and balance.
  * Walk on a treadmill to measure your maximum fitness while wearing a mask to analyze your oxygen use.
  * Blood and urine tests and a heart ultrasound.
  * Questionnaires & activity measures.
  Group assignment for 12 weeks:
  -Exercise classes & activity guidance: Twice-weekly class that focuses on exercises that are similar to daily activities, such as walking and carrying objects. Obtain customized information and education to help you exercise and follow a low salt diet.
  Follow-up:
  -Monthly phone calls during the 12 week follow up period.
  Arms: Functional circuit training and lifestyle counseling
Behavioral: Health education and independent walking — Tests are performed at the beginning, and repeated after 12 and 24 weeks.
  * Measure general fitness levels such as walking, strength and balance.
  * Walk on a treadmill to measure your maximum fitness while wearing a mask to analyze your oxygen use.
  * Blood and urine tests and a heart ultrasound.
  * Questionnaires & activity measures.
  Group assignment for 12 weeks:
  -Health education and walking: Weekly health education classes covering general topics related to heart failure, like medications, diet and exercise. Receive a pedometer for an at-home walking program.
  Follow-up:
  -No follow up support
  Arms: Health education and independent walking

SUMMARY:
Diastolic heart failure is now being recognized as a key form of heart failure in older people. The focus of this research is to study ways to improve and maintain physical activity and functioning. This knowledge may improve the health and well-being in people with diastolic heart failure.

DETAILED DESCRIPTION:
The purpose of this project is to better understand how endurance and fatigue relate to performing daily activities and how we might better improve endurance and reduce fatigue through an exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and over
* Evidence of diastolic dysfunction on echocardiogram
* Normal Left Ventricular Function (LVEF≥50%)
* Heart Failure-NYHA Class II/III
* Able and willing to participate in exercise program
* Able to come to Ann Arbor Michigan for testing

Exclusion Criteria:

* Regularly exercising(30 minute per day, 3 times per week)
* Orthopedic or musculoskeletal condition that limits weight bearing
* Uncontrolled atrial fibrillation
* History of heart valve replacement
* Unstable or serious medical condition (ie. on dialysis, oxygen; severe anemia, uncontrolled blood pressure or coronary artery disease)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
6 minute walk | Baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Mobility Research Center, Ann Arbor, Michigan, United States